CLINICAL TRIAL: NCT01814228
Title: Efficacy of Transcatheter Ablation Using Anatomic Approach of Ganglionated Plexi Located in the Right Atrium to Prevent Neuromediated Cardioinhibitory Syncope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, MD, FESC, Policlinico Casilino ASL RMB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Casilino0001, 0002
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Neuromediated Cardioinhibitory Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- right atrium ganglionated plexi transcatheter ablation (Experimental): right atrium ganglionated plexi transcatheter ablation
  Interventions: Procedure: transcatheter ablation of ganglionated plexi in right atrium

INTERVENTIONS:
Procedure: transcatheter ablation of ganglionated plexi in right atrium

SUMMARY:
Cardioinhibitory neurocardiogenic syncope (CNS) or vasovagal syncope, is the most frequent aetiology of syncope in young people without apparent cardiac or neurological pathology. It is usually caused by inappropriately trigger-activated cardiac reflex which finally precipitates asystole, sinus bradycardia, or atrioventricular (AV) block [1]. Despite young patients affected by CNS have an excellent prognosis when electro-structural heart diseases are excluded [2], their quality of life may be seriously affected by recurrent episodes [2, 3]. Cardiac pacing might help to control symptoms and therefore is considered in patients aged more than 40 years old with recurrent episodes and documented cardioinhibitory response [1, 4]. In young individuals, the role of cardiac pacing is dubious due to predicted frequent device substitutions and adverse ventricular remodeling over time. Recently, radiofrequency (RF) biatrial ablation of ganglionated plexi (GP) has showed promising results in the short and long-term treatment of reflex syncope, functional atrioventricular block, or sinus node dysfunction [5, 6]. Nonetheless, strong evidences are emerging about efficacy of transcatheter ablation limited to ganglionated plexi in the right atrium with the possibility to avoid side-effects related to left-sided procedures [6]

Aim of study

To evaluate in a large cohort of patients effectiveness and safety of gangliar transcatheter ablation in the right atrium to obtain atrial denervation and prevent CNS.

Study population and methods

Twenty consecutive patients affected by cardioinhibitory neurocardiogenic syncope will be enrolled in the study.

Inclusion criteria:

* age between 18 and 60 years
* 3 syncopal episodes at least of likely CNS in the previous 2 years
* marked cardioinhibitory response to HUT or documented asystolic pauses at internal loop recorder registration [7].

Cardioinhibition will be considered as elicitation of asystolic pause (sinus arrest or AV block) ≥ 3 seconds associated to syncope or ≥ 6 seconds and related presyncope.

Exclusion criteria:

* documented myocardial and/or valvular abnormalities on 2D echocardiogram (ejection fraction lower than 50%)
* documented tachyarrhythmias as possible causes of symptoms
* channelopathies (Brugada syndrome, LQT or SQT syndrome)
* ventricular preexcitation
* symptomatic orthostatic hypotension diagnosed by standing blood pressure measurement
* pregnancy in women
* previous cardiac pacemaker implantation.

After obtaining informed consent patients will undergo to basal electrophysiological study (EPS) to record AH interval, HV interval, Wenckebach cycle length, sinus node recovery time (SNRT) and correct sinus node recovery time (cSNRT); the same parameters will be recorded immediately after ablation. Following basal EPS an accurate (200 valid points at least) electroanatomic right atrium mapping (CARTO 3™ Biosense Webster, Inc) will be performed and subsequently radiofrequency delivered at right atrial anatomic sites where the underlying presence of ganglionated plexi (GPs) clusters was regarded as highly probable, on the basis of anatomical studies [8-11]: the supero-posterior area (superior right atrial GP, adjacent to the junction of the superior vena cava and the posterior surface of RA), the middleposterior area (posterior right atrial GP, posterior surface of the RA adjacent the interatrial groove), the infero-posterior area (inferior right GP placed between the inferior vena cava, coronary sinus ostium, and near the atrioventricular groove). Transcatheter ablation will be performed using an 8mm-tip catheter (Biosence-Webster Navistar DS 8mm) or an irrigated 4 mm-tip catheter with force control system (Biosence Webster Smarttouch). Ablation will be performed until complete elimination of local atrial electrical activity. Response to radiofrequencies delivery will be considered successful in case of asystolic pause or cardiac cycle lengthening of 30% (compared to basal cycle) at least. To prolong RF delivery despite asystolic response, a quadripolar catheter will be positioned in right ventricle to backup stimulation. To avoid phrenic nerve injury, high amplitude stimulation will be performed just before radiofrequency delivery to the superior right atrial GP.

HRV analysis will be performed on admission, at 2 hour after ablation and patients discharge. The HRV analysis will include the following parameters: mean, maximal and minimal heart rate, SDNN (standard deviation of Normal-Normal), RMSSD (root mean square successive difference), pNN50 (percentage of differences between adjacent N-N intervals that are >50 msec), LF (low frequency), HF (high frequency).

Moreover, an HUT and an HRV analysis will be performed at 1, 3, 6 and 12 months after ablation procedure during the follow up.

ELIGIBILITY:
Twenty consecutive patients affected by cardioinhibitory neurocardiogenic syncope will be enrolled in the study.

Inclusion criteria:

* age between 18 and 60 years
* 3 syncopal episodes at least of likely CNS in the previous 2 years
* marked cardioinhibitory response to HUT or documented asystolic pauses at internal loop recorder registration [7].

Cardioinhibition will be considered as elicitation of asystolic pause (sinus arrest or AV block) ≥ 3 seconds associated to syncope or ≥ 6 seconds and related presyncope.

Exclusion criteria:

* documented myocardial and/or valvular abnormalities on 2D echocardiogram (ejection fraction lower than 50%)
* documented tachyarrhythmias as possible causes of symptoms
* channelopathies (Brugada syndrome, LQT or SQT syndrome)
* ventricular preexcitation
* symptomatic orthostatic hypotension diagnosed by standing blood pressure measurement
* pregnancy in women
* previous cardiac pacemaker implantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
neuromediated cardioinhibitory syncope recurrence | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Casilino, Rome, Lazio, Italy